CLINICAL TRIAL: NCT00693732
Title: Validation of Surrogate Measures in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: NMRC, Singapore (Unknown)
Responsible Party: Principal Investigator, Medicine, Medicine, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: D/06/264
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1, IBS patients (Active Comparator)
  Interventions: Drug: Escitalopram treatment; Behavioral: Quantitative sensory testing
- 2,Healthy controls (Experimental)
  Interventions: Drug: Escitalopram treatment; Behavioral: Quantitative sensory testing

INTERVENTIONS:
Drug: Escitalopram treatment — On study inclusion at Visit 2, patients will be successively randomised using a computer generated randomisation list to either placebo or escitalopram (Lundbeck Export A/S, Singapore) 10mg given at bedtime in the first 2 weeks, followed by 20mg in the next 6 weeks. The treatments will be identical in appearance and will be administered in double-blind fashion. Treatment with any anticoagulants, antidiabetics, antimigraine drugs, antispasmodics, analgesics, psychoactive agents including antidepressants, Zelmac®, TCM or acupuncture for IBS and any drugs affecting nociception as judged by investigator are prohibited during the entire study.
  Other Names: Lexapro
Behavioral: Quantitative sensory testing — Rectal Distention Stimulation

SUMMARY:
Visceral and somatic hypersensitivity as evidence of central sensory sensitization occur in the majority of Irritable Bowel Syndrome (IBS) patients. We recently demonstrated abnormal endogenous pain modulation as a cause of the sensitization in IBS and identified the underlying dysfunctional neuromatrix using functional MR-imaging (fMRI). Endogenous pain mechanisms regulate, fine-tune and integrate sensory and homeostatic, including neuroendocrine, immune and autonomic nervous system processes. Specific measures of sensitization and endogenous pain modulation correlate with clinical measures of somatic and neuropathic pain, suggesting usefulness as surrogate markers for clinical pain outcomes. Validation of experimental measures as surrogate markers in IBS would provide a considerable advance in pathophysiological and therapeutic research in this pharmacoeconomically burdensome disease.

ELIGIBILITY:
Inclusion Criteria:

IBS patients:

* One hundred fifty male and female IBS patients (Rome III criteria), aged 18 to 70 years, recruited from primary and secondary care via advertisements and referral networks.
* Minimum IBS symptom rating of 75 in IBS severity scoring system (IBS-SSS) in last two weeks.
* IBS discomfort or pain must have been patient's most prominent symptom.
* A minimum of 40 patients each IBS-constipated (IBS-C) and IBS-diarrhoeic (IBS-D) (Rome III) to be included.
* Patients must have been off all IBS and analgesic medication and any drugs potentially influencing sensory function for at least two weeks before study start.

Healthy controls:

* Fifteen healthy controls aged 18 to 70 years without any gastrointestinal pathology or history of significant abdominal pain, bowel disorders, bloating or discomfort during the last 3 months.

Exclusion Criteria:

Exclusion criteria for both IBS patients and healthy controls:

* Organic gastrointestinal or other significant systemic disease, including cardiovascular, psychiatric, neurological and endocrine diseases, as judged by investigator
* Chronic or acute pain, except related to other functional syndromes (functional dyspepsia, chronic pelvic pain, fibromyalgia, migrane)
* Bowel resections (except appendectomy)
* Multiple abdominal operations, excluding hysterectomy
* History of brain disease or brain surgery
* Ongoing treatment with any anticoagulants, antidiabetics, antimigraine drugs, antispasmodics, analgesics, psychoactive agents including antidepressants, Zelmac®, TCM or acupuncture for IBS and any drugs affecting nociception as judged by investigator within last 14 days
* Treatment with any investigational drug during the preceding 30 days
* Pregnancy or lactation.
* Claustrophobia
* Metal implants in body (fMRI exclusion criterion)
* No written informed consent obtained from subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To correlate clinical measures of IBS activity with experimental measures of central sensitisation and endogenous pain modulation | 3 years
  1. To correlate clinical measures of IBS activity with experimental measures of central sensitisation and endogenous pain modulation over the course of six months
  2. To correlate changes in brain and brainstem activation patterns in a subgroup of 15 patients and 15 controls by functional MRI with clinical IBS activity, symptom and pain scores, experimental measures of central sensitisation and endogenous pain modulation over the course of six months.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - NUH, Singapore, Singapore
  - National University Hospital, Singapore